CLINICAL TRIAL: NCT05511298
Title: Empowering Students Project
Status: Recruiting | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: 90ZD0017
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Relationship, Social

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Relationship Smarts Combo — The intervention is a combination of Mind Matters, Relationship Smarts 4.0, and Money Habitudes curricula, developed by the Dibble Institute

SUMMARY:
The Empowering Students Project is an evaluation of the effectiveness of a psychoeducational program for adolescents, intended to help youth build healthy relationship skills while supporting positive socioemotional development and promoting successful transition to young adulthood.

DETAILED DESCRIPTION:
Participants complete measures of the primary outcomes immediately prior to beginning the intervention and again immediately after completion of the program. Analyses will examine within-person change from pre-test to post-test.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Max Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Students who are enrolled in schools (or other programs) that opt to offer the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 1332 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Change in Relationship Quality | Baseline: Immediately prior to the first workshop session; Follow-up: Immediately following the last workshop session (ranging from ~4-8 weeks in between time points, depending on how the workshop is delivered)
  For participants who are in a relationship: Ten items, scored on a 5-point scale and averaged, for a possible range of 1-5. Sample item: "My boyfriend/girlfriend and I talk about the things that really matter."
  For participants who are not in a relationship: Six items, scored on a 4-point scale and averaged, for a possible range of 1-4. Sample item: "I have the skills needed for a lasting, stable romantic relationship."
  Higher scores reflect better outcomes.
Change in Communication Skills | Baseline: Immediately prior to the first workshop session; Follow-up: Immediately following the last workshop session (ranging from ~4-8 weeks in between time points, depending on how the workshop is delivered)
  For participants who are in a relationship: Six items, scored on a 5-point scale and averaged, for a possible range of 1-5. Sample item: "How often do you discuss your disagreements?"
  For participants who are not in a relationship: Five items, scored on a 4-point scale and averaged, for a possible range of 1-4. Sample item: "Listening to another person's opinion during a disagreement."
  Higher scores reflect better outcomes.
Change in Knowledge About Healthy Relationships | Baseline: Immediately prior to the first workshop session; Follow-up: Immediately following the last workshop session (ranging from ~4-8 weeks in between time points, depending on how the workshop is delivered)
  Eight items, scored on a 4-point scale and averaged, for a possible range of 1-4. Sample item: "In a healthy relationship, how important is it that couples do not cheat on each other?"
  Higher scores reflect better outcomes.
Knowledge about Intimate Partner Violence | Baseline: Immediately prior to the first workshop session; Follow-up: Immediately following the last workshop session (ranging from ~4-8 weeks in between time points, depending on how the workshop is delivered)
  Four items, scored on a 4-point scale and averaged, for a possible range of 1-4. Sample item: "It's okay to stay in a relationship even if you're afraid of your boyfriend/girlfriend."
  Higher scores reflect better outcomes.
Change in Increased Knowledge, Skills, and Confidence | Baseline: Immediately prior to the first workshop session; Follow-up: Immediately following the last workshop session (ranging from ~4-8 weeks in between time points, depending on how the workshop is delivered)
  Three items, scored on a 4-point scale and averaged, for a possible range of 1-4. Sample item: "I have learned new skills in this program that I plan to use in my relationships."
  Higher scores reflect better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- The Parenting Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT05511298/SAP_000.pdf